CLINICAL TRIAL: NCT02270424
Title: A Multi-center, Randomized, Double-blind, Controlled Study to Evaluate the Effectiveness of on Severe / Very Severe COPD Patients
Brief Title: Effect of Traditional Chinese Medicine on Outcomes in Patients With Severe / Very Severe COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for severe COPD
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Medicine, Chinese Traditional; Humans; Treatment Outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional medicine+ placebo TCM (Experimental): Patients in this group will be given conventional medicine, Salmeterol / fluticasone based on the classes of medications recommended by 2011 GOLD and Chinese Treatment Guidelines for COPD, and three placebo TCM treatment, which are which are placebo Bufeijianpi granule, placebo Bufeiyishen granule and placebo Yiqizishen granule corresponding to the three traditional Chinese syndromes in sequence, which are syndrome of deficiency of pulmono-splenic qi, syndrome of insufficiency of qi of the lung and kidney, syndrome of insufficiency of qi and yin of the lung and kidney.
  Interventions: Drug: Salmeterol / fluticasone (Seretide®); Drug: Placebo Bufeijianpi granule; Drug: Placebo Bufeiyishen granule; Drug: Placebo Yiqizishen granule
- conventional medicine+ TCM (Experimental): Patients in this group will receive Salmeterol / fluticasone based on the classes of medications recommended by 2011 GOLD and Chinese Treatment Guidelines for COPD, and three types of TCM treatment, which are Bufeijianpi granule, Bufeiyishen granule and Yiqizishen granule. A herbal extract twice daily for 52 weeks for lower dosage. The three granules are corresponding to the three traditional Chinese syndromes in sequence, which are syndrome of deficiency of pulmono-splenic qi, syndrome of insufficiency of qi of the lung and kidney, syndrome of insufficiency of qi and yin of the lung and kidney.
  Interventions: Drug: Salmeterol / fluticasone (Seretide®); Drug: Bufeijianpi granule; Drug: Bufeiyishen granule; Drug: Yiqizishen granule

INTERVENTIONS:
Drug: Salmeterol / fluticasone (Seretide®) — According to the revised 2013 GOLD, Salmeterol / fluticasone was used to severe and very severe COPD patients for 52weeks: Salmeterol / fluticasone (Seretide®, GlaxoSmithKline), 50/500 μg / dose, 60 inhalations. 50/500 μg each time, twice daily.
Drug: Bufeijianpi granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of deficiency of pulmono-splenic qi will be given Bufeijianpi granule, twice daily for 52 weeks for lower dosage.
  Arms: conventional medicine+ TCM
Drug: Bufeiyishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi of the lung and kidney will be given Bufeiyishen granule, twice daily for 52 weeks for lower dosage.
  Arms: conventional medicine+ TCM
Drug: Yiqizishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi and yin of the lung and kidney will be given Yiqizishen granule granule, twice daily for 52 weeks for lower dosage.
  Arms: conventional medicine+ TCM
Drug: Placebo Bufeijianpi granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of deficiency of pulmono-splenic qi will be given placebo Bufeijianpi granule, twice daily for 52 weeks for lower dosage.
  Arms: Conventional medicine+ placebo TCM
Drug: Placebo Bufeiyishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi of the lung and kidney will be given placebo Bufeiyishen granule, twice daily for 52 weeks for lower dosage.
  Arms: Conventional medicine+ placebo TCM
Drug: Placebo Yiqizishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi and yin of the lung and kidney will be given placebo Yiqizishen granule granule, twice daily for 52 weeks for lower dosage.
  Arms: Conventional medicine+ placebo TCM

SUMMARY:
The aim of this study is to compare the effectiveness of two treatments for severe / very severe COPD patients: one, conventional medicine based on 2013 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines; the other, TCM treatments and conventional medicine, which have been evaluated and have certain effect.

DETAILED DESCRIPTION:
Patients with severe or very severe COPD are more likely to suffer repeated exacerbations and more rapidly declining lung function generating increased risk of death and time to a COPD related hospitalization. Although many therapies exist and are being developed to relieve symptoms and reduce mortality in COPD, most have only been studied in moderate to very severe COPD. There are few clinical trials to compare therapeutic alternatives in severe and very sever COPD. Furthermore, some randomized controlled trials on comprehensive Traditional Chinese medicine (TCM) interventions, especially based on the TCM patterns, have been the certain evidence for showing definite effect for COPD patients. In addition, a study about the effect of TCM on outcomes in mild and moderate COPD patients has been in progress and will be carried out in December 2014 (NCT01486186). Hence, corresponding to the mild to moderate COPD patients, The this study aims to evaluate the effectiveness of TCM on severe / very severe COPD patients.

This is a multi-center, randomized, double-blind, controlled study to evaluate the effectiveness of TCM on severe / very Severe COPD patients. Following a 14 day run-in period, approximately 564 subjects will be randomly assigned to conventional medicine treatment group, TCM and conventional medicine treatment group for 52 weeks. After the 52 weeks treatment period, subjects in two treatments arms will follow-up 52 weeks. The primary outcome measure is the frequency of exacerbations. The secondary efficacy measures include all-cause mortality, FEV1, dyspnea (MMRC), exercise capacity( 6MWD), quality of life ( CAT, SF-36 and COPD-PRO), and effectiveness satisfaction with treatment(ESQ-COPD) . Safety will be assessed through the collection of adverse events. There will be a total of 9 study visits (baseline, the 13, 26, 39 and 52 weeks of the treatment, the 13, 26, 39 and 52 weeks of follow-up).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of severe to very severe COPD.
* medically stable
* Age between 40 and 80 years.
* Syndrome differentiation belongs to syndrome of deficiency of pulmonosplenic qi, syndrome of insufficiency of qi of the lung and kidney, syndrome of insufficiency of qi and yin of the lung and kidney.
* with a two-week wash-out period prior to randomization
* Without participations in other interventional trials in the previous one month.
* With the informed consent signed.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Current respiratory disorders other than COPD (e.g., bronchiectasis, bronchial asthma, tuberculosis, lung fibrosis, pulmonary thromboembolic, diffuse panbronchiolitis).
* Complicated with a neuromuscular disorder, which affected the respiration.
* Complicated with heart failure (NYHA Class III or IV),or myocardial infarction within six months ,or unstable hemodynamics.
* Complicated with malignancy, congenital or acquired immune deficiency.
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation).
* Participating in other trials or allergic to the used medicine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The frequency of exacerbation | Change from Baseline in the frequency of exacerbation at the week13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase

SECONDARY OUTCOMES:
Mortality | 52 Weeks of the treatment phase and the 52 Weeks of the followup phase
  The mortality of COPD and all-cause mortality will be calculated.
Forced expiratory volume in one second | Change from Baseline in the one second (FEV1) at the week13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase.
  FEV1 is the amount of air that can be exhaled in one second. A positive change from baseline in FEV1 indicates improvement in lung function.
Dyspnea | Change from Baseline in MMRC at the week13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase
  Using Modified Medical Research Council ( MMRC) scale to assess a patient's level of dyspnea. The MMRC scale is a simple grading system that scored from 0 (less severe) to 4 (severe).
6 Minutes Walking Distance Test ( 6MWD) | Change from Baseline in the 6MWD at the week 13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase.
Quality of life | Change from Baseline in the CAT, SF-36 and COPD-PRO at the week 13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase.
  Using three instruments, COPD Assessment Test ( CAT) , Short Form 36-Item Health Survey (SF-36) and patient reported outcome for chronic obstructive pulmonary disease (COPD-PRO), to asses the impact of COPD on a person's life, and how this changes over time.
Effectiveness satisfaction with treatment | Change from Baseline in the ESQ-COPD at the week 13, 26, 39 and 52 of the treatment phase, the week 13, 26, 39 and 52 of the followup phase.
  Using the effectiveness satisfaction questionnaire of chronic obstructive pulmonary disease (ESQ-COPD) to evaluate COPD patients' satisfaction with their treatment over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine

REFERENCES:
- [Derived] Li J, Xie Y, Wang M, Li S, Yu X, Zhang N, Zhu Z, Zhang W, Feng J, Sun Z, Lin L, Sun Z, Zhang H, Yu X. Effect of traditional Chinese medicine combined with conventional Western medicine for patients with severe/very severe chronic obstructive pulmonary disease: a multi-center, randomized, double-blind, controlled study. Chin Med. 2025 May 20;20(1):66. doi: 10.1186/s13020-025-01117-x. PMID 40394700